CLINICAL TRIAL: NCT04162444
Title: Short-term and Midterm Results of the Aortic Valve Reconstruction With Autopericardium in Children
Brief Title: Results of the Aortic Valve Reconstruction in Children
Status: Recruiting | Type: Observational
Sponsor: National Medical Research Center for Children's Health, Russian Federation (Other Government)
Responsible Party: Sponsor
Other Study IDs: 16072019
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Aortic Valve Insufficiency
Keywords: Aortic Valve Insufficiency/surgery; Aortic Valve/surgery; Child; Reconstructive Surgical Procedures/methods; Cardiac Surgical Procedures; Hemodynamics; Pericardium/transplantation; Transplantation, Autologous; Treatment Outcome; Heart Valve Prosthesis Implantation
MeSH Terms: conditions — Aortic Valve Insufficiency | interventions — Physical Examination; Echocardiography, Transesophageal; Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: We will study safety, clinical and hemodynamic efficacy of the method of the aortic valve reconstruction with autopericardium in children with aortic valve disease.
  Interventions: Diagnostic Test: Physical examination; Diagnostic Test: The Ross Classification for Heart Failure in Children; Diagnostic Test: The Aristotle score; Other: Assessment of administered specific therapy; Diagnostic Test: Multispiral computed tomography/3D echocardiography; Diagnostic Test: Transthoracic and transesophageal echocardiography; Diagnostic Test: 12-lead electrocardiogram

INTERVENTIONS:
Diagnostic Test: Physical examination — A physical examination is a routine screening procedure used to investigate a patient's symptoms or complaints. It consists of a series of questions regarding patient medical history followed by an examination of the symptoms to determine the correct diagnosis and treatment plan.
  Other Names: Medical examination; Clinical examination
Diagnostic Test: The Ross Classification for Heart Failure in Children — The assessment is performed by pediatric cardiologist according to the classic Ross scale. One of the 4 classes of chronic heart failure is registered.
  Other Names: Assessment of heart failure according to Ross scale
Diagnostic Test: The Aristotle score — Surgical risks will be assessed by the ARISTOTLE score developed specially for the task. The calculation will be performed online, available from http://www.aristotleinstitute.org.
  Other Names: Assessment of surgical risks according to the ARISTOTLE score
Other: Assessment of administered specific therapy — The data will be registered as groups of administered medicines:
  * Antiplatelet agents
  * Loop diuretics
  * Potassium-sparing diuretics
  * Angiotensin-converting enzyme inhibitors
Diagnostic Test: Multispiral computed tomography/3D echocardiography — All patients enrolled in the study should be routinely examined with multispiral computed tomography (MS-CT) or 3D-echo before surgery and 3 years later. As a result, a 3D aortic root reconstruction will be made to assess its size and anatomy and subsequently build a 3D soft model for surgery imitation.
  At the study onset, we plan to perform MS-CT, then 3D-echo. If the correlation resulting from 3D-echo and the actual sizes will be high, the isolated 3D-echo will be preferred in the future.
  If none of the methods is available, the patients will not be enrolled in the study.
  The following data will be registered for further analysis:
  * Perimeter of the aortic valve
  * Diameter of the aortic valve at sinuses level
  * Height of the aortic sinuses
  * Morphology of the aortic valve
  Other Names: MS-CT/3D-echo
Diagnostic Test: Transthoracic and transesophageal echocardiography — Transthoracic echocardiography is carried out at baseline, at discharge and then annually. It is performed in order to assess the contractile function of the heart and hemodynamic characteristics of the aortic valve and its autopericardium graft.
  Transesophageal echocardiography is carried out directly after the withdrawal of the artificial circulation when performing augmentation of the aortic valve with autopericardium in order to asses hemodynamic characteristics of the aortic neo-valve.
Diagnostic Test: 12-lead electrocardiogram — Registering 12-lead electrocardiogram (ECG) is used as a tool for assessment of the regularity of the heart rhythm as well as screening and predictive tool for assessment of fibrosis and hypertrophy processes in the myocardium. The following data will be registered:
  * Heart rate
  * Sinus rhythm (yes/no)
  * Positive R wave in leads V5-6
  * Angle α less than 0
  * Presence/absence of abnormal Q wave
  * Presence/absence of ST-segment depression in precordial leads
  Other Names: 12-lead ECG

SUMMARY:
Aortic valve disease counts up to 5% of cases of congenital heart disease being one of the most common congenital malformations of the cardiovascular system. This disease requires replacement of the damaged valve which in itself is not a trivial task to complete in children as there is still no available best practice for valve replacement. Today, the following alternative variants are performed in children: mechanical aortic prosthesis, xenografts, allografts, and pulmonary autograft (Ross procedure) and each has its potential advantages and disadvantages.

Mechanical aortic prostheses require lifelong anticoagulation therapy and repeated surgeries to replace mechanical valves during child growth. Available xenografts in children also has suboptimal results not only because of absence of growth potential, but also due to development of degenerative changes in biological tissue of the graft leaflets. Allograft tissues are exposed to rapid biodegradation in the recipient body and thus requiring repeated surgeries associated with higher difficulty, high risk of hemorrhages, and injury of the coronary injuries. Ross procedure was proposed as theoretically the most evidence-based reconstruction of the aortic valve in children. Even successfully performed Ross operation transforms one-valve disorder into two-valve disease.

The accumulation of knowledge on the anatomy of the aortic root and improvement of surgical techniques led to the development of new methods for reconstruction of the valve function. The technique is widely applied in adult cardiac surgery, uses glutaraldehyde-treated autopericardium for augmentation of the leaflets. Absence of foreign material provides no need for anticoagulation therapy. Potentially, reconstruction of the aortic valve with autopericardium can be widely used in children.

Aim is to study safety, clinical and hemodynamic efficacy of the method of the aortic valve reconstruction with autopericardium in children with aortic valve disease. Patients aged 29 days to 12 years will be included into the study. The data according to the protocol of the study will be assessed at the stage of inclusion, during the surgery, in 30 days after the surgery, and in 1, 2, and 3 years after the surgery. Data about all the patients included into the research will be analyzed in order to study the endpoints and achieve the research aim.

DETAILED DESCRIPTION:
Aortic valve disease amounts to approximately 5% of the total number of cases of congenital heart disease, thus being one of the most common congenital malformations of the cardiovascular system. This disease requires replacement of the damaged valve, which in itself is not a trivial task to complete in children as there is still no available perfect option for valve replacement. Today, the following alternative variants for the aortic valve reconstruction in children are known: mechanical aortic prosthesis, xenografts, allografts and pulmonary autograft (Ross procedure); each of the above-mentioned variants has its potential advantages and disadvantages.

Mechanical aortic prostheses are widely available, including in small sizes (16 and 18 mm) appropriate for young children. However, the available sizes still do not allow to perform the surgical reconstruction in children of the first year of life. Besides these patients need lifelong anticoagulation therapy and necessity for repeated surgeries in order to replace mechanical valves with a child's growth.

Available xenografts have various types but usually, their sizes begin from 19 mm which does not fit for the majority of young children. Aortic xenografts are characterized by low risk of thromboembolism complications and do not require lifelong antithrombotic therapy. However, application of these grafts in children also has suboptimal results not only because of the absence of growth potential but also due to the development of degenerative changes in biological tissue of the graft leaflets.

Allografts are characterized by perfect hemodynamic parameters which are similar to the native healthy aortic valve. Risk of thromboembolic complications in implantation of allografts is very low, so there is no need for anticoagulation therapy. As in xenografts, allograft tissues are exposed to rapid biodegradation in the recipient body with the following development of obstruction or insufficiency and thus requiring a repeat operation. Implantation of allografts is associated with higher difficulty and high risk of hemorrhages and injury of the coronary injuries.

Ross procedure was proposed as theoretically the most justified choice for reconstruction of the aortic valve in children. As a conduit for reconstruction of the aortic valve the host's intact native pulmonary valve - autograft - is used; and the pulmonary valve is usually replaced by xenograft. Even successfully performed Ross operation, according to some authors, resolves the problem of the aortic valve only for a while; moreover, it causes another problem with the pulmonary valve, thus transforming one-valve disorder into two-valve disease.

The accumulation of knowledge on the anatomy of the aortic root and improvement of surgical techniques has led to the development of new methods for reconstruction of the valve function. The experience of various options for interventions on the aortic valve leaflet gained in adult cardiac surgery allowed to consider such interventions as an alternative method to valve reconstruction in children. About ten years ago, Professor Shigeyuki Ozaki brought the reconstruction of the aortic valve with the patient's own tissues to a completely new technological level. This technique includes the use of glutaraldehyde-treated autopericardium for augmentation of the leaflets; the reproducibility of the method was significantly increased due to usage of the template sets and special tools for the measurement of the native valve. Since no foreign material is used, there is no need for anticoagulation therapy after such intervention, which the authors of the method referred to as the valve reconstruction, not implantation of the graft. Potentially, reconstruction of the aortic valve with autopericardium can be widely used in children. In this population of patients, the various variants of the leaflets dysmorphogenesis are much more common, a wide range of morphological diversity of structure with inadequate hemodynamics can be found: monocuspid, bicuspid and pseudobicuspid valves; which does not allow to perform the valve reconstruction by restoring the original anatomy.

The normal anatomy of the aortic valve assumes three-valve structure, and most augmentation techniques suppose formation of tricuspid anatomy. At the same time, there is an alternative variant of hemodynamically adequate valve structure in the human body - bicuspid anatomy of the venous valves in the vena cava inferior system. Theoretical calculations obtained through computer simulation show that the neo-valve formed by three artificial leaflets will retain its locking function with increasing the diameter of the fibrous ring only by 8%. At the same time, the bicuspid valve with an increased height of the leaflets is able to maintain the shut-off function with an increase in the diameter of the fibrous ring by 67%.

The aim is to study safety, clinical and hemodynamic efficacy of the method of the aortic valve reconstruction with autopericardium in children with aortic valve disease. Primary endpoints: patient's death due to various causes during the first 30 days after the surgery. Secondary endpoints for efficacy assessment: аreedom from repeated surgeries on the aortic valve; mean gradient at the aortic valve over 40 mmHg; аortic insufficiency over 2 degree; effective area of the neo-aortic valve less than 1.0 cm2/m2 Secondary endpoint for safety assessment: acute disorders of cerebral circulation within the first 30 days after the surgery; hemorrhage needing revision surgery; acute kidney injury, stages 2 or 3, including the necessity for renal replacement therapy; acute coronary syndrome; dysfunction of the neo-valve requiring repeated surgery.

Patients aged from 29 days to 12 years old with dysfunction of the native aortic valve with and without manifestations, with indications for the aortic valve reconstruction, and without concomitant supravalvular and subvalvular aortic stenosis and major congenital heart diseases, will be included into the study. The study design is planned to be prospective, cohort, single-center, observational. In total 40 patients will be included into the study. The data according to the protocol of the study will be assessed at the stage of inclusion, during the surgery, in 30 days after the surgery, and in 1, 2, and 3 years after the surgery. Data about all the patients included in the research will be analyzed in order to study the endpoints and achieve the research aim.

The first report on safety of the operation will be published when all the patients included in the study are carried out the procedure of augmentation of the aortic valve with autopericardium and all of them are examined within 30 days after the surgery. A report about the efficacy of the operation within the first year after the performed surgery of augmentation of the aortic valve with autopericardium; it will be published after all the patients included in the study are examined at the control visit in one year after the surgery. Report about clinical and hemodynamic efficacy of the operation within three years after the performed reconstruction of the aortic valve with autopericarduim; it will be published after all the patients included in the study are examined in three years after the surgery. Final report on the study will be published when for all patients included in the study all the follow-up periods are completed, or patients are excluded from the study due to other causes.

For compensation for the lost quantitative or qualitative data, statistical methods will not be applied. If there is a lack in patient's data due to any causes, such a patient will be excluded from this block of analysis. A number of patients included in each analysis will be represented in the report, so readers could themselves assess the influence of the lost data on the published result.

ELIGIBILITY:
Inclusion Criteria:

* Age from 29 days to 12 years
* Patient's official caregivers have to sign the informed consent after they are thoroughly explained the meaning of the study, its protocol and timelines.
* Patients with manifestations, with mean gradient at the aortic valve >40 mmHg with normal left ventricular ejection fraction (LVEF), or patients with manifestations with the mean gradient < 40 mmHg with decreased LVEF, or patients with manifestations with severe aortic insufficiency, or patients without manifestations, but with decreased LVEF with aortic insufficiency, or patients with concomitant moderate aortic insufficiency and moderate aortic stenosis with manifestations.
* Aortic Z-score over -1,5
* Absence of subvalvular and supravalvular aortic stenosis
* Absence of intracardiac malformations requiring correction, except for septal defects

Non-inclusion criteria:

* Known hypersensitivity to aspirin, heparin, nitinol, intravenous contrast or contradictions to their administration due to other causes.
* Previous replacement of the aortic valve with mechanical or xenografts.
* Confirmed active sepsis or endocarditis.
* Hypoplasia of the fibrous ring of the aortic valve with Z score under -1,5.
* Life expectancy less than 3 years due to concomitant diseases.
* Participation in another clinical research.
* Indications for urgent surgery.
* Intracardiac malformations requiring momentary surgical correction.
* Geographical instability of a patient and his/her official caregivers, complicating significantly the constant contact during the study

Exclusion Criteria:

• Refusal of patient's caregivers to participate further in the study.

Ages: 29 Days to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will enroll the participants from the patients of the the Department of Cardiac Surgery with dysfunction of the native aortic valve with and without manifestations, with indications for the aortic valve reconstruction, and without concomitant supravalvular and subvalvular aortic stenosis and major congenital heart diseases.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-02-18 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Death Rate | From baseline till 1 month after the surgery
  Patient's death due to various causes during the first 30 days after the surgery.

SECONDARY OUTCOMES:
Number of Participants with Repeat Aortic Valve Surgery | During the 5-6 years of the follow-up period since the surgery
  We will observe if a patient had an emergency for the repeat surgery on the aortic valve
Number of Participants with Aortic Valve Mean Gradient over 40 mmHg | During the 5-6 years of the follow-up period since the surgery
  We will register the cases when the mean gradient at the aortic valve will exceed 40 mmHg
Number of Participants with Aortic Insufficiency Stage 2-4 | During the 5-6 years of the follow-up period since the surgery
  We will register the cases when the patients will be diagnosed with aortic insufficiency Stage 2-4
Neo-aortic valve effective area less than 1.0 cm2/m2 | During the 5-6 years of the follow-up period since the surgery
  We will register the cases when the effective area of the neo-aortic valve will be less than 1.0 cm2/m2
Number of Participants with Hemorrhage requiring surgery | During the 5-6 years of the follow-up period since the surgery
  We will register the patients diagnosed with a hemorrhage requiring surgery
Number of Participants with Acute Disorders of Cerebral Circulation | During the first 30 days after the surgery
  We will register the patients with acute disorders of cerebral circulation after the surgery
Number of Participants with Acute Kidney Injury Stages 2 or 3 | During the 5-6 years of the follow-up period since the surgery
  We will register the patients with acute kidney injury Stages 2 or 3, including those requiring renal replacement therapy
Number of Participants withAcute Coronary Syndrome | During the 5-6 years of the follow-up period since the surgery
  We will register the patients diagnosed with acute coronary syndrome
Number of Participants with Dysfunction of the Neo-valve Requiring Repeat Intervention | During the 5-6 years of the follow-up period since the surgery
  We will register the cases when patients are diagnosed with dysfunction of the neo-valve after the surgery and require repeated operation

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry V. Ryabtsev, PhD, Principal Investigator — National Research Center of Children's Health
Locations (1):
- National Medical Research Center of Children's Health, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made available partially upon a request.
Supporting Information: Study Protocol
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: IPD will be shared upon a request.

REFERENCES:
- [Result] Salomon NW, Stinson EB, Oyer P, Copeland JG, Shumway NE. Operative treatment of congenital aortic stenosis. Ann Thorac Surg. 1978 Nov;26(5):452-60. doi: 10.1016/s0003-4975(10)62925-6. PMID 753159
- [Result] Brown JW, Ruzmetov M, Vijay P, Rodefeld MD, Turrentine MW. Surgery for aortic stenosis in children: a 40-year experience. Ann Thorac Surg. 2003 Nov;76(5):1398-411. doi: 10.1016/s0003-4975(03)01027-0. PMID 14602258
- [Result] Karamlou T, Jang K, Williams WG, Caldarone CA, Van Arsdell G, Coles JG, McCrindle BW. Outcomes and associated risk factors for aortic valve replacement in 160 children: a competing-risks analysis. Circulation. 2005 Nov 29;112(22):3462-9. doi: 10.1161/CIRCULATIONAHA.105.541649. PMID 16316968
- [Result] Alsoufi B. Aortic valve replacement in children: Options and outcomes. J Saudi Heart Assoc. 2014 Jan;26(1):33-41. doi: 10.1016/j.jsha.2013.11.003. Epub 2013 Nov 13. PMID 24578598
- [Result] Alsoufi B, Al-Halees Z, Manlhiot C, McCrindle BW, Al-Ahmadi M, Sallehuddin A, Canver CC, Bulbul Z, Joufan M, Fadel B. Mechanical valves versus the Ross procedure for aortic valve replacement in children: propensity-adjusted comparison of long-term outcomes. J Thorac Cardiovasc Surg. 2009 Feb;137(2):362-370.e9. doi: 10.1016/j.jtcvs.2008.10.010. PMID 19185153
- [Result] Ruzmetov M, Vijay P, Rodefeld MD, Turrentine MW, Brown JW. Evolution of aortic valve replacement in children: a single center experience. Int J Cardiol. 2006 Nov 10;113(2):194-200. doi: 10.1016/j.ijcard.2005.11.011. Epub 2006 Jan 10. PMID 16376439
- [Result] Alsoufi B, Manlhiot C, McCrindle BW, Canver CC, Sallehuddin A, Al-Oufi S, Joufan M, Al-Halees Z. Aortic and mitral valve replacement in children: is there any role for biologic and bioprosthetic substitutes? Eur J Cardiothorac Surg. 2009 Jul;36(1):84-90; discussion 90. doi: 10.1016/j.ejcts.2009.02.048. Epub 2009 Apr 14. PMID 19369085
- [Result] Polimenakos AC, Sathanandam S, Elzein C, Barth MJ, Higgins RS, Ilbawi MN. Aortic cusp extension valvuloplasty with or without tricuspidization in children and adolescents: long-term results and freedom from aortic valve replacement. J Thorac Cardiovasc Surg. 2010 Apr;139(4):933-41; discussion 941. doi: 10.1016/j.jtcvs.2009.12.015. PMID 20304137
- [Result] Lupinetti FM, Duncan BW, Lewin M, Dyamenahalli U, Rosenthal GL. Comparison of autograft and allograft aortic valve replacement in children. J Thorac Cardiovasc Surg. 2003 Jul;126(1):240-6. doi: 10.1016/s0022-5223(03)00041-2. PMID 12878961
- [Result] Solowiejczyk DE, Bourlon F, Apfel HD, Hordof AJ, Hsu DT, Crabtree G, Galantowicz M, Gersony WM, Quaegebeur JM. Serial echocardiographic measurements of the pulmonary autograft in the aortic valve position after the Ross operation in a pediatric population using normal pulmonary artery dimensions as the reference standard. Am J Cardiol. 2000 May 1;85(9):1119-23. doi: 10.1016/s0002-9149(00)00707-4. PMID 10781763
- [Result] Elkins RC, Knott-Craig CJ, Ward KE, McCue C, Lane MM. Pulmonary autograft in children: realized growth potential. Ann Thorac Surg. 1994 Jun;57(6):1387-93; discussion 1393-4. doi: 10.1016/0003-4975(94)90089-2. PMID 8010778
- [Result] Solymar L, Sudow G, Holmgren D. Increase in size of the pulmonary autograft after the Ross operation in children: growth or dilation? J Thorac Cardiovasc Surg. 2000 Jan;119(1):4-9. doi: 10.1016/s0022-5223(00)70211-x. PMID 10612754
- [Result] Simon P, Aschauer C, Moidl R, Marx M, Keznickl FP, Eigenbauer E, Wolner E, Wollenek G. Growth of the pulmonary autograft after the Ross operation in childhood. Eur J Cardiothorac Surg. 2001 Feb;19(2):118-21. doi: 10.1016/s1010-7940(00)00638-2. PMID 11167098
- [Result] Hraska V, Krajci M, Haun Ch, Ntalakoura K, Razek V, Lacour-Gayet F, Weil J, Reichenspurner H. Ross and Ross-Konno procedure in children and adolescents: mid-term results. Eur J Cardiothorac Surg. 2004 May;25(5):742-7. doi: 10.1016/j.ejcts.2004.01.009. PMID 15082276
- [Result] Elkins RC, Thompson DM, Lane MM, Elkins CC, Peyton MD. Ross operation: 16-year experience. J Thorac Cardiovasc Surg. 2008 Sep;136(3):623-30, 630.e1-5. doi: 10.1016/j.jtcvs.2008.02.080. PMID 18805263
- [Result] Alsoufi B, Al-Halees Z, Manlhiot C, McCrindle BW, Kandeel M, Al-Joufan M, Kalloghlian A, Fadel B, Canver CC. Superior results following the Ross procedure in patients with congenital heart disease. J Heart Valve Dis. 2010 May;19(3):269-77; discussion 278. PMID 20583388
- [Result] Hazekamp MG, Grotenhuis HB, Schoof PH, Rijlaarsdam ME, Ottenkamp J, Dion RA. Results of the Ross operation in a pediatric population. Eur J Cardiothorac Surg. 2005 Jun;27(6):975-9. doi: 10.1016/j.ejcts.2005.01.018. PMID 15896604
- [Result] Takkenberg JJ, Klieverik LM, Schoof PH, van Suylen RJ, van Herwerden LA, Zondervan PE, Roos-Hesselink JW, Eijkemans MJ, Yacoub MH, Bogers AJ. The Ross procedure: a systematic review and meta-analysis. Circulation. 2009 Jan 20;119(2):222-8. doi: 10.1161/CIRCULATIONAHA.107.726349. Epub 2008 Dec 31. PMID 19118260
- [Result] Alsoufi B, Manlhiot C, Fadel B, Al-Ahmadi M, Tamim M, McCrindle BW, Canver CC, Al-Halees Z. The Ross procedure in children: preoperative haemodynamic manifestation has significant effect on late autograft re-operation. Eur J Cardiothorac Surg. 2010 Nov;38(5):547-55. doi: 10.1016/j.ejcts.2010.03.025. Epub 2010 Apr 21. PMID 20409726
- [Result] Woods RK, Pasquali SK, Jacobs ML, Austin EH, Jacobs JP, Krolikowski M, Mitchell ME, Pizarro C, Tweddell JS. Aortic valve replacement in neonates and infants: an analysis of the Society of Thoracic Surgeons Congenital Heart Surgery Database. J Thorac Cardiovasc Surg. 2012 Nov;144(5):1084-89. doi: 10.1016/j.jtcvs.2012.07.060. Epub 2012 Aug 24. PMID 22921819
- [Result] Shinkawa T, Bove EL, Hirsch JC, Devaney EJ, Ohye RG. Intermediate-term results of the Ross procedure in neonates and infants. Ann Thorac Surg. 2010 Jun;89(6):1827-32; discussion 1832. doi: 10.1016/j.athoracsur.2010.02.107. PMID 20494035
- [Result] Hickey EJ, Yeh T Jr, Jacobs JP, Caldarone CA, Tchervenkov CI, McCrindle BW, Lacour-Gayet F, Pizarro C. Ross and Yasui operations for complex biventricular repair in infants with critical left ventricular outflow tract obstruction. Eur J Cardiothorac Surg. 2010 Feb;37(2):279-88. doi: 10.1016/j.ejcts.2009.06.060. Epub 2009 Sep 17. PMID 19762251
- [Result] Alsoufi B, Al-Halees Z, Manlhiot C, Awan A, Al-Ahmadi M, McCrindle BW, Al-Joufan M, Canver CC. Intermediate results following complex biventricular repair of left ventricular outflow tract obstruction in neonates and infants. Eur J Cardiothorac Surg. 2010 Oct;38(4):431-8. doi: 10.1016/j.ejcts.2010.02.035. Epub 2010 Apr 10. PMID 20382029
- [Result] David TE. Aortic Valve Replacement in Children and Young Adults. J Am Coll Cardiol. 2016 Jun 21;67(24):2871-3. doi: 10.1016/j.jacc.2016.04.023. No abstract available. PMID 27311526
- [Result] Duran CM, Gometza B, Kumar N, Gallo R, Martin-Duran R. Aortic valve replacement with freehand autologous pericardium. J Thorac Cardiovasc Surg. 1995 Aug;110(2):511-6. doi: 10.1016/S0022-5223(95)70248-2. PMID 7637369
- [Result] Duran CM, Gallo R, Kumar N. Aortic valve replacement with autologous pericardium: surgical technique. J Card Surg. 1995 Jan;10(1):1-9. doi: 10.1111/j.1540-8191.1995.tb00582.x. PMID 7696782
- [Result] Ozaki S, Kawase I, Yamashita H, Uchida S, Nozawa Y, Matsuyama T, Takatoh M, Hagiwara S. Aortic valve reconstruction using self-developed aortic valve plasty system in aortic valve disease. Interact Cardiovasc Thorac Surg. 2011 Apr;12(4):550-3. doi: 10.1510/icvts.2010.253682. Epub 2011 Jan 27. PMID 21273254
- [Result] Ozaki S, Kawase I, Yamashita H, Uchida S, Nozawa Y, Takatoh M, Hagiwara S. A total of 404 cases of aortic valve reconstruction with glutaraldehyde-treated autologous pericardium. J Thorac Cardiovasc Surg. 2014 Jan;147(1):301-6. doi: 10.1016/j.jtcvs.2012.11.012. Epub 2012 Dec 8. PMID 23228404
- [Result] Zhang HF, Ye M, Yan XG, Chen G, Tao QL, Jia B. Application of a Simplified Hand-Sewn Trileaflet Valved Conduit in Right Ventricular Outflow Tract Reconstruction as an Alternative for Bovine Jugular Vein Graft: Single-Center Experience. Artif Organs. 2018 Jan;42(1):41-48. doi: 10.1111/aor.12968. Epub 2017 Oct 2. PMID 28971487
- [Result] Hosseinpour AR, Gonzalez-Calle A, Adsuar-Gomez A, Santos-deSoto J. A simple method of aortic valve reconstruction with fixed pericardium in children. Interact Cardiovasc Thorac Surg. 2013 May;16(5):695-7. doi: 10.1093/icvts/ivs547. Epub 2013 Jan 23. PMID 23343835
- [Result] Hammer PE, Roberts EG, Emani SM, Del Nido PJ. Surgical reconstruction of semilunar valves in the growing child: Should we mimic the venous valve? A simulation study. J Thorac Cardiovasc Surg. 2017 Feb;153(2):389-396. doi: 10.1016/j.jtcvs.2016.08.019. Epub 2016 Aug 31. PMID 27665220
- [Result] Dashkevich A, Blanke P, Siepe M, Pache G, Langer M, Schlensak C, Beyersdorf F. Preoperative assessment of aortic annulus dimensions: comparison of noninvasive and intraoperative measurement. Ann Thorac Surg. 2011 Mar;91(3):709-14. doi: 10.1016/j.athoracsur.2010.09.038. PMID 21352983
- [Result] Ross RD. The Ross classification for heart failure in children after 25 years: a review and an age-stratified revision. Pediatr Cardiol. 2012 Dec;33(8):1295-300. doi: 10.1007/s00246-012-0306-8. Epub 2012 Apr 5. PMID 22476605
- [Result] Lacour-Gayet F, Clarke D, Jacobs J, Comas J, Daebritz S, Daenen W, Gaynor W, Hamilton L, Jacobs M, Maruszsewski B, Pozzi M, Spray T, Stellin G, Tchervenkov C, Mavroudis And C; Aristotle Committee. The Aristotle score: a complexity-adjusted method to evaluate surgical results. Eur J Cardiothorac Surg. 2004 Jun;25(6):911-24. doi: 10.1016/j.ejcts.2004.03.027. PMID 15144988
- [Result] Bigi S, Fischer U, Wehrli E, Mattle HP, Boltshauser E, Burki S, Jeannet PY, Fluss J, Weber P, Nedeltchev K, El-Koussy M, Steinlin M, Arnold M. Acute ischemic stroke in children versus young adults. Ann Neurol. 2011 Aug;70(2):245-54. doi: 10.1002/ana.22427. PMID 21823153
- [Result] RANKIN J. Cerebral vascular accidents in patients over the age of 60. II. Prognosis. Scott Med J. 1957 May;2(5):200-15. doi: 10.1177/003693305700200504. No abstract available. PMID 13432835
- See also: Dhand NK, Khatkar MS. (2014). Statulator: an online statistical calculator. Sample Size Calculator for Estimating a Single Proportion. Accessed 15 March 2019 — http://statulator.com/SampleSize/ss1P.html